CLINICAL TRIAL: NCT00466882
Title: Issues Related to the Use of the INAMED LAPBAND SYSTEM to Reduce BMI's in Obese Renal Failure Patients Needing Renal Transplantation: A Pilot Study
Brief Title: Use of the INAMED LAPBAND System to Reduce BMI's in Obese Renal Failure Patients
Status: Withdrawn | Type: Observational
Why Stopped: No patients were enrolled.
Sponsor: Summa Health System (Other)
Responsible Party: Principal Investigator, John Zografakis, Staff Surgeon, Summa Health System
Other Study IDs: INAMED
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Renal Failure; Obesity
Keywords: obese; renal failure; renal transplant candidate; Hemodialysis BMI between 36 and 42
MeSH Terms: conditions — Renal Insufficiency; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Inamed Lap-Band System: The LAPBAND is positioned laparoscopically around the stomach and requires an overnight hospitalization and an upper GI swallow the next morning. The device can be gradually adjusted to increase stomach constriction by the physician in an office setting so that the patient loses approximately 1-2 pounds per week over two years.
  Interventions: Device: Inamed Lap-Band System

INTERVENTIONS:
Device: Inamed Lap-Band System — Patient's will be seen in the physician's office one week post surgery and once a month thereafter. The device can be gradually adjusted by the insertion of a needle into the port and saline is added or removed to inflate or deflate the LAPBAND. This can be conducted in the physician's office setting to enable the patient to lose 1-2 pounds per week over two years.

SUMMARY:
The purpose of this study is to assess the use of this Lap-Band system for the purpose of promoting weight loss in renal failure patients who do not qualify as transplant candidates because of excessive BMI's

DETAILED DESCRIPTION:
The concern of transplant surgeons is that obese patients with high BMI's are more likely to experience post-transplantation complications than age-matched recipients [1]. Nevertheless, the Summa transplant list contains numerous patients with renal failure that have BMI's above 35. These patients are not considered to be "active" transplant candidates because of their obesity and are not eligible to receive a kidney transplant. Dr. Lal counsels these patients that they must lose weight in order to be considered active candidates for transplantation.

Weight loss for obese patients in renal failure is difficult. These patients must undergo hemodialysis three times weekly. Most of these patients do not, or physically cannot, engage in exercise activities. Many of these patients are burdened psychologically, and further behavioral responsibilities related to weight loss may overstress them. Repetitive diets or behavioral therapy in morbidly obese patients prior to transplantation have had disappointing results [2]. Likewise, pharmacological management of obesity in these patients is largely unsuccessful. Noradrenergic appetite suppressants must be restricted because of stimulatory side-effects. Serotonergic agents have cardiovascular and pulmonary complications. Thermogenic agents are minimally effective [2].

The INAMED LAPBAND SYSTEM is an FDA-approved, surgically-placed device marketed to facilitate weight reduction in obese individuals. The LAPBAND is positioned laparoscopically around the stomach and requires an overnight hospitalization and an upper GI swallow the next morning. The device can be gradually adjusted to increase stomach constriction by the physician in an office setting so that the patient loses approximately 1-2 pounds per week over two years. These adjustments are performed on average 4-5 times during the first year and twice during the second year.

The purpose of this pilot study is to assess the utility of the LAPBAND in facilitating weight loss in obese renal failure patients awaiting transplantation and to document issues related to its use in these patients. The hope is that the LAPBAND will facilitate enough weight loss to reduce the patient's BMI to 35 or below after placement of the LAPBAND. If the patient reaches the intended goal of BMI of 35, they will be placed on the active renal transplant list and will be eligible for transplantation.

A secondary goal of this research is to follow those patients who successfully reach BMI's of 35 or less who are subsequently transplanted to determine any untoward effects of the LAPBAND upon transplantation success

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* Hemodialysis patient with BMI between 36 and 42

Exclusion Criteria:

* Patients undergoing peritoneal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with renal failure that have BMI's above 35 that would be a candidate for renal transplant if their BMI were 35 or less
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-10-17 (Actual); Primary Completion 2010-11 (Estimated); Study Completion 2011-01-24 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 2 years
  Assess weight loss after surgery

SECONDARY OUTCOMES:
Transplantation Success | 2 years
  Assess possible effects of weight loss surgery on transplantation success

CONTACTS AND LOCATIONS:
Overall Officials: John Zografakis, MD, Principal Investigator — Summa Health System; Tanamay Lal, MD, Principal Investigator — Summa Health System
Locations (1):
- Summa Health System, Akron, Ohio, United States